CLINICAL TRIAL: NCT05420376
Title: Prospective Comparison of Whole Mesh and Split Mesh Use in Patient Groups Undergoing Laparoscopic Inguinal Hernia Repair
Brief Title: Comparison of Whole Mesh and Split Mesh Use in Laparoscopic Inguinal Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erol Aydın, General Surgeon, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 569874
Record Dates: First submitted 2022-05-20; First posted 2022-06-15 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Hernia, Inguinal
Keywords: Laparoscopic Inguinal Hernia; Laparoscopic Hernia; Whole Mesh; Split Mesh; TAP; TEPP; Inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Mesh (Active Comparator): For the patients in the first group, the whole patch will be laid on the area without being fixed.
  Interventions: Procedure: Split Mesh
- Split Mesh (Active Comparator): The patients in the second group will be given a patch of the same size, but partially divided horizontally and wrapped around the spermatic cord.
  Interventions: Procedure: Split Mesh

INTERVENTIONS:
Procedure: Split Mesh — TEP repair of inguinal hernias using either split or whole mesh
  Other Names: Whole mesh

SUMMARY:
At least 80 patients who will undergo laparoscopic inguinal hernia repair surgery will be randomized into 2 groups. For the patients in the first group, the whole mesh will be laid on the area without being fixed. The patients in the second group will be given a mesh of the same size, but partially divided horizontally and wrapped around the spermatic cord. Demographic data of patients in both groups, quality of life data(Carolinas Comfort Scale) at postoperative 1st, 7th, 30th, 3rd and 6th months, postoperative pain (VAS values), clinical seroma rate, recurrence and other complications will be monitored. When the desired number of patients and follow-up period are reached, the data in the 2 groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Clinical or/and radiological diagnosed primary inguinal hernia
* TEP or TAPP surgical methods

Exclusion Criteria:

* Recurrent hernias
* Patients with previous groin operations on same side
* Pregnant women
* Patients who did not accept to participate in the study
* ASA score of 3 or higher,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2023-05-16 (Estimated); Study Completion 2023-06-16 (Estimated)

PRIMARY OUTCOMES:
Carolinas Comfort Scale values | 6 month
  Differences in postoperative pain and quality of life(Carolinas Comfort Scale at first month) in patients who use whole meshes and those who use split meshes.
Recurrence rates | 6 month
  Differences in recurrence rates in patients who use whole meshes and those who use split meshes.

SECONDARY OUTCOMES:
Recurrence rates | 6 month
  Difference in recurrence rates at 6 months in patients who use whole meshes and those who use split meshes.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided